CLINICAL TRIAL: NCT03382626
Title: Transcranial Direct Current Stimulation and Computer-based Training for the Rehabilitation of Cognitive Function in Traumatic Brain Injury: a Randomized Controlled Trial
Brief Title: Transcranial Direct Current Stimulation and Computer-based Training for the Traumatic Brain Injury Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Renato Anghinah, Doctor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 71391917000000068
Record Dates: First submitted 2017-12-04; First posted 2017-12-26 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Transcranial Direct Current Stimulation; Computer-assisted training; Cognitive training; Cognitive function; Executive function; Working memory; Attention
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Prospective, double-blind, randomized, parallel, controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS plus Computer-assisted training (Active Comparator): Patients will receive 10 sessions of active anodal tDCS on the left prefrontal cortex dorsolateral (F3 area using International 10-20 system for electroencephalogram (EEG) electrode placement) plus Computer-assisted cognitive training (games to improve working memory, attention, and executive function).
  Interventions: Device: anodal tDCS; Device: Computer-assisted training
- tDCS sham plus Computer-assisted training (Sham Comparator): Patients will receive 10 sessions of sham anodal tDCS on the left prefrontal cortex dorsolateral plus Computer-assisted cognitive training (games to improve working memory, attention and executive function).
  Interventions: Device: Computer-assisted training; Device: sham tDCS

INTERVENTIONS:
Device: anodal tDCS — Anodal tDCS will be applied on the left prefrontal cortex dorsolateral (F3 area using International 10-20 system for EEG electrode placement) with the following parameters: electrode size of 25-35 cm², 2mA, 0.057 mA/cm² and duration of 20 minutes. The cathode will be placed over the supra-orbital region.
  Arms: tDCS plus Computer-assisted training
Device: Computer-assisted training — The computer-assisted cognitive training will consist of games with visual and auditory stimuli to improve working memory, attention, and executive function. The games will be Genius and Labyrinth games, reaction time and timing-coincident.
Device: sham tDCS — Sham tDCS will be applied with the same parameters and electrode placement of active anodal tDCS. However, the current flow will be interrupted by the device after few seconds.
  Arms: tDCS sham plus Computer-assisted training

SUMMARY:
Traumatic Brain Injury (TBI) is a serious public health problem due to its high mortality and morbidity rates, mainly affecting young adult males. Aggression to the prefrontal cortex, caused by an external physical force, responsible for anatomical injury and/or functional impairment, causes cognitive deficits with important consequences for the individual affected by the trauma and their caregivers. Therefore, rehabilitation is of utmost importance. The increase in pre-frontal cortical activation through training, activity-dependent stimulation and neuroplasticity, especially in the dorsolateral prefrontal cortex (DLPFC) is related to better performance in functional memory. In this context, Transcranial Direct Current Stimulation (tDCS), intended to drive neuroplastic changes in the brain, has been widely used to bring benefits to the cognitive function of individuals affected by various neurological conditions, including TBI by promoting neuroplasticity for critically involved cortical areas in the performance of tasks, culminating in cognitive benefits. In addition, studies have shown greater benefits when the technique is combined with cognitive training. Therefore, the objective of this parallel, randomized, double-blind, placebo-controlled clinical trial is to investigate the effect of tDCS applied on the dorsolateral prefrontal cortex and virtual reality cognitive training alone or in association with tDCS on cognitive function of individuals with severe chronic TBI.

ELIGIBILITY:
Inclusion Criteria:

* Chronic TBI (≥ 12 months)
* Severe TBI (Glasgow ≤ 8, loss of consciousness > 24 hours, post-traumatic amnesia > 1 week)
* Working memory, attention or executive deficit
* Score in Mini Mental State Examination according the cut-off point (i.e, 13 to illiterates individuals, 18 to low and medium schooling and 26 to high schooling).

Exclusion Criteria:

* Individuals unable to perform the activities proposed in the study protocol (e.g. physical deficits, lack of collaboration, aphasia, accuses, amaurosis)
* Mid or extensive cranial defects
* Titanium cranial prosthesis
* Extensive cranial prosthesis located on the dorsal prefrontal cortex
* Metallic devices implanted in the brain
* Psychotic disorders
* Recent history of alcoholism or use of drugs
* Neurological diseases (e.g Parkinson, Stroke, Alzheimer).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-02-19 (Actual); Primary Completion 2018-11-30 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline working memory at 10 days of intervention (scale assessment) | We will apply these instruments at T0 (baseline time), T2 (at end of all sessions, i.e 10 days after the first session) and T3 (i.e after 1 month of follow-up time).
  Will be performed throughWechsler Adult Intelligence Scale IV (Digit span, Letter-Number Sequencing and Arithmetic subtests). These subtests evaluates the working memory and attention. The Digit span involves a forward and a backward recitation condition. The maximum score is 30 points, where higher score indicates better the performance. Letter-Number sequencing involves a combination of numbers and letters that must be recited.The maximum scores is 21 points, where higher scores shows better performance. The Arithmetic subtest is formed by some calculations must be solved without the aid of paper and pen. The maximum score is 22 points in which higher scores indicates better performance. The score of each subtest will be considered separately for characterization of the working memory. In addition, The sum of the weighted individual scores in each subtest will be calculated for the Working Memory Index.
Change from baseline working memory at 10 days of intervention (computer-based assessment) | We will apply these instruments at T0 (baseline time), T1 (one day after the first session), T2 (at end of all sessions, ie 10 days after the first session) and T3 (i.e after 1 month of follow-up time).
  This assessment will occur through the Genius game, which will evaluate the performance in the unit of measure of execution time (i.e. seconds) of the task.
Change from baseline executive function at 10 days of intervention (scale assessment) | We will apply these instruments at T0 (baseline time), T2 (at end of all sessions, ie 10 days after the first session) and T3 (i.e after 1 month of follow-up time).
  This assessment will occur through the Trail Making Test A and B, which provides information on visual search, scanning, speed of processing, mental flexibility, and executive functions. It requires the subject to connect encircled numbers randomly arranged on a page (Part A) and encircled numbers and letters in alternating order (Part B). Scoring is expressed in time in seconds required for completion of each of the two parts of the test. Scoring is expressed in terms of the time in seconds required for completion of each of the two parts of the test, on which the shorter the time to complete the task the better the performance (i.e part A < 180 s and part B < 300 s).
Change from baseline attention and executive function at 10 days of intervention (scale assessment) | We will apply these instruments at T0 (baseline time), T2 (at end of all sessions, ie 10 days after the first session) and T3 (i.e after 1 month of follow-up time).
  This assessment will occur through the Stroop Color and Word Test, which assesses the ease with which a person can maintain a goal in mind and suppress the habitual response in favor of a less familiar one (i.e selective attention and cognitive flexibility). Both the time to complete and the number of errors. In addition, the interference effect is determined by calculating the extra time required to name colors in the interference task in comparison to the time required to name colors in the control task.
Change from baseline processing speed at 10 days of intervention (scale assessment) | We will apply these instruments at T0 (baseline time), T2 (at end of all sessions, ie 10 days after the first session) and T3 (i.e after 1 month of follow-up time).
  This assessment will occur through the Code Search subtest (WAIS), which as evaluates the processing speed to complete a card with number and symbols that must be related to a correct execution of the test. The score is formulated based on correct answers. The maximum score is 133 points. The higher scores are related to better performance.

SECONDARY OUTCOMES:
Change from baseline processing speed at 10 days of intervention (computer-based assessment) | We will apply these instruments at T0 (baseline time), T1 (one day after the first session), T2 (at end of all sessions, ie 10 days after the first session) and T3 (i.e after 1 month of follow-up time).
  This assessment will occur through the following instruments: Reaction time game and Timing Coincident game. These computer games measure the score in the unit of measure of time, where the lower the execution time the better the performance (i.e processing speed).
Change from baseline reasoning and planning at 10 days of intervention (computer-based assessment) | We will apply these instruments at T0 (baseline time), T1 (one day after the first session), T2 (at end of all sessions, ie 10 days after the first session) and T3 (i.e after 1 month of follow-up time).
  This evaluation will be performed through the maze game, in which performance is measured by the task execution time. Thus, the shorter the execution time, the better the cognitive performance.
Change from baseline quality of life at 10 days of intervention | We will apply the QOLIBRI at T0 (baseline time), T2 (at end of all sessions, ie 10 days after the first session) and T3 (i.e after 1 month of follow-up time).
  This assessment will occur through Quality of Life After Brain Injury (QOLIBRI) scale, which is a comprehensive questionnaire with 37 items covering six dimensions (cognition, self, daily life and autonomy, social relationships, emotion and physical problems). The scale means are converted to the 0-100 scale by subtracting 1 from the mean and then multiplying by 25. This produces scale scores which have a lowest possible value of 0 (worst possible quality of life) and a maximum value of 100 (best possible quality of life).
Change from baseline depression at 10 days of intervention | We will apply the BDI at T0 (baseline time), T2 (at end of all sessions, ie 10 days after the first session) and and T3 (i.e after 1 month of follow-up time).
  This assessment will occur through Beck Depression Inventory (BDI), which is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.

OTHER OUTCOMES:
Adverse effects assessment | We will apply the AEQ at end of each sessions of anodal tDCS (i.e one by day during 10 days)
  This assessment will occur through Adverse effects Questionaire (AEQ), which is an instrument developed for directed and self-rated adverse effects assessment. Therefore, it has no scores.
Sociodemographic and Neurological assessment | We will apply this questionnaire only at T0 (baseline time)
  This assessment will occur through Sociodemographic and Neurological Questionnaire, built on Common Data Elements for TBI -NINDS for directed evaluation of sociodemographic aspects; data collection of brain trauma, such as: history of trauma, cause, mechanism of action, type of TB, affected brain area, degree of trauma, time of trauma, etc .; pre-existing diseases, comorbidities, signs and symptoms and medications in use.
Mental state examination assessment | We will apply this questionnaire only at T0 (baseline time)
  This assessment will occur through Mini-mental state examination, wich evaluates cognitive function. The maximum score is 30 points, consisting of two domains: test for vocal responses, orientation, memory and attention (maximum of 21 points); and test for naming ability, verbal and written commands, spontaneous writing of a sentence and copying of a complex polygon (maximum of nine points).

CONTACTS AND LOCATIONS:
Locations (1):
- Ambulatório de Reabilitação Cognitiva do Hospital das Clínicas da Universidade de São Paulo, São Paulo, Brazil